CLINICAL TRIAL: NCT03660735
Title: The PIP Study- Pre- IVF Immune Profiling Study
Brief Title: The PIP Study - Pre- IVF Immune Profiling Study
Acronym: PIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Finox Biotech (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13399
Record Dates: First submitted 2018-07-09; First posted 2018-09-07 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Sub-fertility; Recurrent Implantation Failure
Keywords: Immune Profiling; Pre-IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Per participant the study will require a maximum of 30ml of blood this will be taken via 3xLiHep 4.5ml vacutainers and 1 x EDTA 4.5ml vacutainer.
  Endometrial biopsy samples will be obtained using an Endocell Disposable endometrial cell sampler. The biopsy tissue will be transferred into 10ml falcon tube containing sterile PBS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Male Factor Subfertility: Participant is undergoing first or second cycle of IVF and ICSI for male factor subfertility
- Recurrent Implantation Failure: Participant is undergoing an IVF cycle to treat subfertility with a history of Recurrent Implantation Failure (RIF).
- Female Subfertility: Participant is undergoing an IVF cycle to treat at least 1 year of subfertility

SUMMARY:
Many IVF clinics offer testing for immune cells in the blood and endometrium as it has been suggested that abnormal levels of these cells can affect fertility or the chance of an IVF cycle working. However, routinely offering these tests remains highly controversial as the scientific evidence behind the tests is not of a high quality. The PIP Study aims to find out how a woman's blood and endometrial immune cells affect the likelihood of an IVF cycle working and whether or not they are different in women with subfertility and implantation failure. This feasibility study aims to find out if it is possible to enrol enough women into the research study. If this is successful, the investigators will then go on to recruit a larger group of women into the main PIP study to enable them to investigate the impact of immune profiling on IVF success in more detail.

DETAILED DESCRIPTION:
Although there are examples of autoimmune associated pregnancy pathology, notably the anti-phospholipid syndrome (1), robust evidence of immune mediated pregnancy failure is limited. However for many years there have been persistent reports of a possible association between 'abnormal' levels of peripheral or endometrial immune cell populations (predominantly NK cells), altered cell function or cytokine production (by NK and T cells) and subfertility, recurrent failed implantation or recurrent miscarriage (2-5). Many fertility clinics offer testing for a variety of peripheral blood immune cell parameters (NK cell numbers, cytotoxicity assays, Tregs, cytokine assays, etc) or endometrial parameters (most commonly NK cell numbers). Furthermore, treatments including corticosteroids, immunoglobulin, intralipids, biologic agents (e.g.: anti-TNFα therapy) are commonly offered to treat 'abnormal' results. The testing and treatment of immune mediated subfertility and implantation failure remains highly controversial for a number of reasons:

1. To date there is little evidence that blood or endometrial immune cell numbers, activation status or function, are associated with either implantation failure or successful IVF treatment (6).
2. There is little evidence in the literature as to normal parameters of endometrial or blood immune cell populations in fertile women. Of note, a recent meta-analysis (6) of blood NK cells describes a total of 106 fertile controls and compares them to 249 women who were either subfertile or had recurrent implantation failure. This is the largest dataset of controls however the 6 included studies vary in how the cells were measured and therefore pooling these data is of limited value. Studies assessing endometrial NK cells comprised only 20 fertile women and 40 subfertile women.
3. The majority of studies compare a pathology (e.g.: Recurrent Implantation Failure (RIF)) with controls but do not have outcome data of the subsequent IVF cycles.
4. It is often argued that blood testing can be of no value as the immune cell populations in the endometrium are phenotypically and functionally different to those in the periphery (7). However the majority of clinical testing is done in blood. There are only a few small studies that compare endometrial and blood parameters in the same patients with no evidence to date that blood NK cells reflect the endometrial NK population.

The evidence above describes the limited data on which routine clinical testing is performed. Added to which, there are no high quality Randomised Controlled Trials showing evidence of benefit for the treatments that are used. In this study the investigators propose to describe in detail normal endometrial and blood immune cell parameters as this has not previously been done in a large population In order to achieve this, women who are undergoing a first cycle or second cycle of IVF for male factor subfertility requiring Intracytoplasmic Sperm injection (ICSI) will be recruited. Those women who go on to have a live birth will be considered to be fertile controls (as their reason for IVF was a male factor and pregnancy was achieved at the first attempt). A sub-group of such participants will be used to describe the normal population (with standard deviations) and to use as a control group to compare to pathologies (RIF and subfertility).

The investigators wish to recruit broadly to the study-250 women overall but they have not defined a recruitment target for each group so that they can, at the end of the feasibility study identify the proportions of the 250 women who fall into each subgroup. Depending on the findings the investigators may need to target specific groups in the main study.

The purpose of the feasibility study is to determine the recruitment rate in the screened population for a larger fully powered study. The investigators will recruit all women under the age of 40 (at time of egg collection) from IVI clinics in the UK and the Wolfson Fertility Centre who are eligible and wish to recruit to the study. Within this population of recruits there will be three specific groups:

1. Women in a first or second cycle of IVF for male factor subfertility requiring ICSI.
2. Women with a history of RIF (using the definition described in (8))
3. Any women with a history of at least 1 year of subfertility.

Inclusion in the study will require women to undertake a single visit to have a blood sample and an endometrial biopsy during the mid-luteal phase of the cycle before IVF treatment. There are minimal risks (besides the small risk of bruising and discomfort) from blood tests. Endometrial biopsy (known clinically as an endometrial 'scratch') is a procedure that is commonly undertaken prior to IVF treatment, as there is evidence that a scratch increases the pregnancy rate in the subsequent IVF cycle (9). Endometrial biopsy causes some discomfort at the time of the procedure but has no significant risks to participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Female, aged 18 years to 39 years at the time of egg collection.
* Participant has an ovulatory cycle of 25-35 days.
* Participant is undergoing:

  * A first or second cycle of IVF and ICSI for male factor subfertility, or
  * An IVF cycle to treat subfertility with a history of RIF, or
  * An IVF cycle to treat at least 1 year of subfertility

We do not plan to target specific numbers in each group. Rather, the numbers that recruit in each group will be assessed at the end of the study and may well influence the design of the main study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Donor egg cycle.
* Age 40 or above at the time of egg collection.
* Ovulatory cycle of <25 or >35 days or evidence of anovulation
* Involved in a interventional research study of any medication that may have an effect on the immune system
* Patient taking oral steroids or other immunomodulatory medication

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants only
Study Population: Participants will be women attending an IVI Midlands, IVI Oxford clinic or the Wolfson Fertility Centre age <40 years who are undertaking an IVF cycle.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment of 250 participants to subgroups relevant to a future larger study | At study completion, this is anticipated to be 3 years.
  Recruitment rate of participants screened eligible for the study
  * of recruits who are undoing a first or second IVF cycle with ICSI for male factor subfertility
  * of recruits with a history of recurrent implantation failure

SECONDARY OUTCOMES:
To describe the normal variation in blood and endometrial immune cell populations in the mid-luteal phase of the menstrual cycle of women in undergoing IVF for a severe male factor subfertility who go on to have a live birth | Blood and endometrial biopsies will be analysed throughout the study (a period of 36 months) but comparison between groups will take place after 3 years, at study completion
  Descriptive data to define the populations of blood and endometrial cells, this will include NK and T cells as well as smaller immune cell populations.
To identify if there are significant differences in endometrial or blood immune cell populations in: Women with a history of Recurrent Implantation Failure Women with a history of subfertility | Blood and endometrial biopsies will be analysed throughout the study (a period of 36 months) but comparison between groups will take place after 3 years, at study completion
  Significant differences in cellular parameters between control group and RIF / subfertility
To identify if there are differences in immune cell parameters between successful and failed cycles | Blood and endometrial biopsies will be analysed throughout the study (a period of 36 months) but comparison between groups will take place after 3 years, at study completion
  Differences in immune cell parameters depending on pregnancy outcome
To identify if there is a relationship between endometrial and peripheral blood immune cell parameters | Blood and endometrial biopsies will be analysed throughout the study (a period of 36 months) but comparison between groups will take place after 3 years, at study completion
  Correlation between endometrial and blood immune cell parameters

OTHER OUTCOMES:
Identify novel differences in the endometrial cellular landscape and cell function in women with recurrent implantation failure and subfertility | Blood and endometrial biopsies will be analysed throughout the study (a period of 36 months) but comparison between groups will take place after 3 years, at study completion
  Comparative studies of endometrial cell phenotype and function, including CyTOF, development in culture, mRNA expression, cytokine levels and response to exogenous factors in control / RIF and subfertility populations

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Granne, DPhil MA MBBS MRCOG, Study Director — University of Oxford
Locations (2):
- United Kingdom (2):
  - Wolfson Fertility Centre, London
  - IVI Oxford, Oxford

REFERENCES:
- [Background] Rai R, Sacks G, Trew G. Natural killer cells and reproductive failure--theory, practice and prejudice. Hum Reprod. 2005 May;20(5):1123-6. doi: 10.1093/humrep/deh804. Epub 2005 Mar 10. PMID 15760961
- [Background] Beer AE, Kwak JY, Ruiz JE. Immunophenotypic profiles of peripheral blood lymphocytes in women with recurrent pregnancy losses and in infertile women with multiple failed in vitro fertilization cycles. Am J Reprod Immunol. 1996 Apr;35(4):376-82. doi: 10.1111/j.1600-0897.1996.tb00497.x. PMID 8739457
- [Background] Kwak-Kim JY, Chung-Bang HS, Ng SC, Ntrivalas EI, Mangubat CP, Beaman KD, Beer AE, Gilman-Sachs A. Increased T helper 1 cytokine responses by circulating T cells are present in women with recurrent pregnancy losses and in infertile women with multiple implantation failures after IVF. Hum Reprod. 2003 Apr;18(4):767-73. doi: 10.1093/humrep/deg156. PMID 12660269
- [Background] Ng SC, Gilman-Sachs A, Thaker P, Beaman KD, Beer AE, Kwak-Kim J. Expression of intracellular Th1 and Th2 cytokines in women with recurrent spontaneous abortion, implantation failures after IVF/ET or normal pregnancy. Am J Reprod Immunol. 2002 Aug;48(2):77-86. doi: 10.1034/j.1600-0897.2002.01105.x. PMID 12389596
- [Background] McGrath E, Ryan EJ, Lynch L, Golden-Mason L, Mooney E, Eogan M, O'Herlihy C, O'Farrelly C. Changes in endometrial natural killer cell expression of CD94, CD158a and CD158b are associated with infertility. Am J Reprod Immunol. 2009 Apr;61(4):265-76. doi: 10.1111/j.1600-0897.2009.00688.x. PMID 19260857
- [Background] Seshadri S, Sunkara SK. Natural killer cells in female infertility and recurrent miscarriage: a systematic review and meta-analysis. Hum Reprod Update. 2014 May-Jun;20(3):429-38. doi: 10.1093/humupd/dmt056. Epub 2013 Nov 27. PMID 24285824
- [Background] Moffett A, Regan L, Braude P. Natural killer cells, miscarriage, and infertility. BMJ. 2004 Nov 27;329(7477):1283-5. doi: 10.1136/bmj.329.7477.1283. PMID 15564263
- [Background] Polanski LT, Baumgarten MN, Quenby S, Brosens J, Campbell BK, Raine-Fenning NJ. What exactly do we mean by 'recurrent implantation failure'? A systematic review and opinion. Reprod Biomed Online. 2014 Apr;28(4):409-23. doi: 10.1016/j.rbmo.2013.12.006. Epub 2014 Jan 17. PMID 24581986
- [Background] Nastri CO, Lensen SF, Gibreel A, Raine-Fenning N, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2015 Mar 22;(3):CD009517. doi: 10.1002/14651858.CD009517.pub3. PMID 25803542